CLINICAL TRIAL: NCT02747082
Title: Antibacterial Effectiveness of Two Root Canal Irrigants in Root-filled Teeth With Infection: A Randomized Clinical Trial
Brief Title: Antibacterial Effectiveness of Two Root Canal Irrigants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Universidade Estácio de Sá (Unknown)
Responsible Party: Principal Investigator, Homan Zandi, DDS, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/364/REK
Record Dates: First submitted 2016-03-21; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Periapical Periodontitis
Keywords: endodontic retreatment; sodium hypochlorite; chlorhexidine; calcium hydroxide; Retreatment
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1% sodium hypochlorite (NaOCl) (Active Comparator): Retreatment of root-filled teeth with infection with 1% NaOCl as irrigation solution.
  Total bacterial counts, Streptococcal species and Enterococcus faecalis species were quantified using qPCR against 16SrRNA before irrigation (S1), after irrigation (S2), and after intracanal medication (S3).
  Interventions: Procedure: Retreatment of root-filled teeth with infection
- 2% chlorhexidine gluconate (CHX) (Active Comparator): Retreatment of root-filled teeth with infection with 2% CHX as irrigation solution.
  Total bacterial counts, Streptococcal species and Enterococcus faecalis species were quantified using qPCR against 16SrRNA before irrigation (S1), after irrigation (S2), and after intracanal medication (S3).
  Interventions: Procedure: Retreatment of root-filled teeth with infection

INTERVENTIONS:
Procedure: Retreatment of root-filled teeth with infection — Root-filled teeth with infection are being treated with either 1% NaOCl or 2% CHX as disinfection irrigation solution.

SUMMARY:
The aim of this randomized clinical trial is to compare the antibacterial effects of 1% sodium hypochlorite (NaOCl) and 2% chlorhexidine gluconate (CHX) during retreatment of teeth with apical periodontitis (AP).

DETAILED DESCRIPTION:
Root canal-treated teeth with AP were randomly distributed in two groups according to the irrigant used. After removal of the previous filling material, bacteriological samples were taken from the canals before (S1) and after chemomechanical preparation using either NaOCl or CHX (S2), and after calcium hydroxide medication for 2-3 weeks (S3). 16S rRNA gene-based real-time qPCR was performed to detect and quantify total bacteria, Streptococcus species and Enterococcus faecalis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of apical periodontitis in a root-filled tooth assessed by radiography.

Exclusion Criteria:

* Presence of gross carious lesions in the diagnosed tooth,
* Presence of fractures involving the periodontium of the diagnosed tooth,
* Presence of periodontal pockets more than 4 mm deep in the diagnosed tooth,
* Diagnosis of diabetes,
* Diagnosis of HIV infection,
* Other immunocompromising disease,
* Antibiotic therapy within the previous 3 months.

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Periapical radiolucency (PAI- and Friedman-scores) | 12 months

SECONDARY OUTCOMES:
Bacterial load assessed by qPCR | 21 days
Pyrosequencing of species found before and after the intervention | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Dag MR Ørstavik, DDS, PhD, Study Chair — Chair of the endodontic department, University of Oslo
Locations (1):
- University of Oslo, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Rocas IN, Siqueira JF Jr. Comparison of the in vivo antimicrobial effectiveness of sodium hypochlorite and chlorhexidine used as root canal irrigants: a molecular microbiology study. J Endod. 2011 Feb;37(2):143-50. doi: 10.1016/j.joen.2010.11.006. PMID 21238793